CLINICAL TRIAL: NCT00371631
Title: Colonizing Neurogenic Bladders With Benign Flora
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B4444-P
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Spinal Cord Injury; Urinary Tract Infection
Keywords: biofilm; clinical trial; Escherichia coli; urinary catheter
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Tract Infections; Escherichia coli Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other): insertion of E. coli coated catheter
  Interventions: Biological: Insertion of urinary catheters coated with E. coli 83972

INTERVENTIONS:
Biological: Insertion of urinary catheters coated with E. coli 83972 — All patients in this pilot study were in the treatment arm, which consisted of receiving a urinary catheter that had been pre-coated with a biofilm of E. coli.

SUMMARY:
The purpose of the research is to determine whether we can get harmless bacteria to live in the bladders of persons with spinal cord injury who practice intermittent bladder catheterization. We will also look at whether having the harmless bacteria in the bladder prevents urinary tract infections from occurring.

DETAILED DESCRIPTION:
The unifying goal of our work is to develop new approaches for the prevention of urinary tract infection (UTI) in persons with spinal cord injury (SCI). Most individuals with SCI have neurogenic bladders, and the resulting urinary stasis and bladder catheterization predispose them to recurrent UTI. Currently few, if any, measures are effective at prevention of UTI in persons with neurogenic bladders.

Bacterial interference, or using benign bacteria to prevent infection with virulent pathogens, may offer a solution to the significant problem of recurrent episodes of UTI in persons with SCI. Two trials in persons with SCI of instilling nonpathogenic Escherichia coli (83972) directly into the bladder demonstrated a strong association between colonization with this non-pathogen and decreased frequency of UTI. However, the successful colonization rate of the direct inoculation method was low (51-62%). Since a urinary catheter-associated biofilm, or bacteria plus extracellular matrix, continually seeds the bladder with bacteria, we proposed to use urinary catheters that had been pre-coated with a biofilm of E. coli 83972 as a means to achieve bladder colonization. Our recently completed pilot (B3248P) demonstrated that insertion of urinary catheters pre-coated with E. coli (83972) was an effective and safe method to achieve bladder colonization with this potentially protective strain. The rate of successful colonization with the E. coli-coated catheters was high (10 of 12 subjects, or 83%). However, this pilot was limited to the subpopulation of SCI veterans who utilize chronic indwelling catheters for bladder drainage.

The current proposal expands upon previous work by widening the range of eligible subjects and by simplifying the colonization protocol. Since an intermittent catheterization program (ICP) is a preferred and more common means of managing neurogenic bladders than chronic catheterization, we now plan to test E. coli 83972-coated catheters in persons with SCI who use ICP for bladder drainage. We hypothesize that short-term use (3 days) of E. coli 83972-coated catheters in persons with SCI practicing ICP will lead to successful colonization (persisting 28 days or more) in the majority of subjects. We will also record subjects' rates of symptomatic UTI while colonized with E. coli 83972 and compare these rates to the subjects' baseline rates in the year prior to study entry. Subjects will be able to remove their study catheters at home and to submit urine samples by mail, so the colonization process will simple and convenient. If successful colonization is achieved in this pilot trial, a larger clinical trial will be designed to test the efficacy of these catheters at preventing UTI in persons with SCI.

ELIGIBILITY:
Inclusion Criteria:

Patients followed at the MEDVAMC who have sustained spinal cord injury > 12 months earlier, suffer from neurogenic bladder, practice intermittent bladder catheterization, and who have had at least 1 symptomatic UTI in the past will be enrolled.

Exclusion Criteria:

Exclusion criteria will include obstructive urolithiasis, indwelling bladder or nephrostomy catheters, supravesical urinary diversion, vesicoureteral reflux, active malignancy, uncontrolled diabetes mellitus, AIDS, requirement for immunosuppressive medication, or current antibiotic therapy. Women of childbearing age must have a negative pregnancy test before enrolling in the study, and they must utilize effective birth control methods during the study and for 3 months after the study is concluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-10; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Trautner, MD, Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (1):
- Michael E DeBakey VA Medical Center, Houston, Texas, United States

REFERENCES:
- [Result] Burns AC, Petersen NJ, Garza A, Arya M, Patterson JE, Naik AD, Trautner BW. Accuracy of a urinary catheter surveillance protocol. Am J Infect Control. 2012 Feb;40(1):55-8. doi: 10.1016/j.ajic.2011.04.006. Epub 2011 Aug 3. PMID 21813209

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: insertion of E. coli coated catheter
  Insertion of urinary catheters coated with E. coli 83972: All patients in this pilot study were in the treatment arm, which consisted of receiving a urinary catheter that had been pre-coated with a biofilm of E. coli.
Period: Overall Study
Arm/Group | Treatment Arm
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 13
Age, Customized [Mean (Full Range); unit: years]
  Age | 56 [37 to 73]
Sex/Gender, Customized [Number; unit: participants]
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
average time since injury [Mean (Full Range); unit: years] | 15 [1.3 to 35]

OUTCOME MEASURES:

1. Primary Outcome: Bladder Colonization
Description: Bladder colonization was defined when (≥102 cfu/ml) of E. coli 83972 was detected in urine cultures for > 3 days after catheter removal.
Time Frame: > 3 days, up to 197 days
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 13
percentage of participants | 62

2. Secondary Outcome: The Rate of Symptomatic UTI While Colonized
Description: Symptomatic UTI was defined as significant bacteriuria (≥105 cfu/ml) and pyuria (>10 WBC/hpf) plus ≥1 of the following signs and symptoms for which no other etiology could be identified: fever (oral temperature >100°F), suprapubic or flank discomfort, bladder spasm, change in voiding habits, increased spasticity, or worsening dysreflexia. The rate of UTI (number) was calculated by dividing the total number of patient days by the total number of UTIs.
Time Frame: 3 years
Measure: Number; unit: UTI/per subject year
Arm/Group | Treatment Arm
Number analyzed (Participants) | 13
UTI/per subject year
  pre-study rate of UTI | 2.27
  post-study rate of UTI | 1.98

ADVERSE EVENTS:
Arm/Group | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=13)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Groin pain (Renal and urinary disorders) | 1 (1)
Dysreflexia (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Lack of placebo control.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes